CLINICAL TRIAL: NCT02433873
Title: Prebiotic Effects of Isomalto-oligosaccharide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Principal Investigator, Cara Frankenfeld, Assistant Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 115796
Record Dates: First submitted 2015-04-25; First posted 2015-05-05 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Microbiota
Keywords: Microbiota; Body weight; Digestive system
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Ingredients that are in the placebo are: high maltose corn syrup (Satin Sweet™), water, and mannitol. Both Supplement A and Supplement B will be compared to this placebo arm.
  Interventions: Dietary Supplement: Isomalto-oligosaccharide
- Supplement A (Experimental): Ingredients that are in the supplement are: isomalto-oligosaccharide, water, mannitol, maltose, glucose, and glycerol. Supplement A and B differ by degrees of polymerization.
  Interventions: Dietary Supplement: Isomalto-oligosaccharide
- Supplement B (Experimental): Ingredients that are in the supplement are: isomalto-oligosaccharide, water, mannitol, maltose, glucose, and glycerol. Supplement A and B differ by degrees of polymerization.
  Interventions: Dietary Supplement: Isomalto-oligosaccharide

INTERVENTIONS:
Dietary Supplement: Isomalto-oligosaccharide — Isomalto-oligosaccharide (IMO) is a non-digestible type of oligosaccharide commonly used as a low-calorie sweetener mixed with a variety of other food and beverage products for the purpose of sweetening.

SUMMARY:
The primary purpose of this study is to evaluate the effect of an IMO nutritional supplement on gut microbiome, gut health, and body weight. Two formulations of the supplement will be evaluated; thus, there will be three study arms: Supplement A, Supplement B, and placebo. Stool samples will be analyzed for bacterial DNA. The gut bacterial DNA, body weight, and gut health data will be compared across supplement and placebo groups.

Primary Aim 1: To evaluate the effect of the IMO supplement on gut bacterial abundance, diversity, and gene function across intervention and placebo groups, and across two doses of the intervention.

Secondary Aim 1: To evaluate the effect of the IMO supplement on gut health across intervention and placebo groups, and across two doses of the intervention.

Secondary Aim 2: To evaluate the effect of the IMO supplement on body weight across intervention and placebo groups, and across two doses of the intervention.

60 subjects, randomized to three arms (20 each: Supplement formula A, Supplement formula B or placebo) will take a daily dose of Supplement A, Supplement B, or placebo for 8 weeks. The supplement is a light syrup liquid. Ingredients that are in the supplement are: isomalto-oligosaccharide, water, mannitol, maltose, glucose, and glycerol. Ingredients that are in the placebo are: high maltose corn syrup (Satin Sweet™), water, and mannitol. Dose will be 500 mg during the first 4 weeks and then 1000 mg for second 4 weeks. Subjects will be instructed to take 500 mg/day of the supplement or placebo the first four weeks and 1000 mg/day of the supplement or placebo for the second four weeks. Subjects will be blinded as to whether they are receiving placebo or supplement. After screening and once enrolled, subject involvement includes visits to George Mason University, being weighed, dropping off stool samples, and completing a survey on gut health. Stool samples will be analyzed for bacterial DNA. The gut bacterial DNA, weight, and gut health data will be compared across supplement and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged 18 to 45 years of age
* In good general health as evidenced by medical history
* Women of reproductive potential must use highly effective contraception
* Body mass index of 25 kg/m2 or higher
* Weigh less than 350 lbs.

Exclusion Criteria:

* History of colon cancer
* History of rheumatoid arthritis
* Active self-reported febrile illness (may enroll after 2-week waiting period following the day that the illness/fever is resolved)
* Taking TNF-alpha inhibitors, COX2 inhibitors, JAK inhibitors
* History of hypothyroidism (with or without treatment)
* History of inflammatory bowel disease (ulcerative colitis and Crohn's disease)
* Type I or Type II diabetes
* History of Parkinson's Disease, Huntington's Disease or Multiple Sclerosis
* History of major depression, bipolar disorder, or schizophrenia
* Pregnant or lactating women
* Currently suffering from migraine headaches (at least one migraine headache in the past 30 days)
* Current use of any prescription or non-prescription weight loss products
* Consumption of more than 2 drinks per day of alcohol
* Tobacco smoker (over ½ pack per week is excluded)
* Marijuana smoker (over once per month is excluded)
* Currently have an eating disorder including anorexia nervosa, bulimia, and/or obsessive compulsive disorders
* Plan to start a new diet or make changes to their current diet during the study
* Diagnosis of Coronary Artery Disease who have had chest pain within the past 2 months
* Diagnosis of Congestive Heart Failure who have had any episodes of shortness of breath within the last 2 months
* History of stroke within the past 1 year
* History of ventricular tachycardia or fibrillation
* History of hypertension that has been difficult to control with medication (based on medical history - e.g. requiring more than 2 medication to achieve control)
* History of seizures in the last 5 years
* Cancer diagnosis in the last 5 years (except non-melanoma skin cancer or in-situ cervical cancer)
* History of bariatric or lapband surgery
* Usual or planned consumption of more than 2 servings per week of yogurt, kombucha, kefir, or kimichi
* Regular use of antibiotics
* Use of antibiotics in the previous 2 weeks
* Current and continued use of prebiotics or probiotics
* Known allergic reactions to components of the study supplement or placebo

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in gut bacterial DNA from baseline, extracted from fecal sample | 4 weeks
Change in gut bacterial DNA from baseline, extracted from fecal sample | 8 Weeks

SECONDARY OUTCOMES:
Body weight change from baseline | Week 4
Change from baseline in self-reported digestive health measured by questionnaire | Week 4
Change from baseline in self-reported digestive health measured by questionnaire | Week 8
Body weight change from baseline | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Cara L Frankenfeld, PhD, Principal Investigator — George Mason University
Locations (1):
- George Mason University, Fairfax, Virginia, United States

REFERENCES:
- [Background] Thitaram SN, Chung CH, Day DF, Hinton A Jr, Bailey JS, Siragusa GR. Isomaltooligosaccharide increases cecal Bifidobacterium population in young broiler chickens. Poult Sci. 2005 Jul;84(7):998-1003. doi: 10.1093/ps/84.7.998. PMID 16050115
- [Background] Chung CH, Day DF. Efficacy of Leuconostoc mesenteroides (ATCC 13146) isomaltooligosaccharides as a poultry prebiotic. Poult Sci. 2004 Aug;83(8):1302-6. doi: 10.1093/ps/83.8.1302. PMID 15339004
- [Background] Chen HL, Lu YH, Lin JJ, Ko LY. Effects of isomalto-oligosaccharides on bowel functions and indicators of nutritional status in constipated elderly men. J Am Coll Nutr. 2001 Feb;20(1):44-9. doi: 10.1080/07315724.2001.10719013. PMID 11294172
- [Background] Wang HF, Lim PS, Kao MD, Chan EC, Lin LC, Wang NP. Use of isomalto-oligosaccharide in the treatment of lipid profiles and constipation in hemodialysis patients. J Ren Nutr. 2001 Apr;11(2):73-9. doi: 10.1016/s1051-2276(01)92591-9. PMID 11295027
- [Background] Yen CH, Tseng YH, Kuo YW, Lee MC, Chen HL. Long-term supplementation of isomalto-oligosaccharides improved colonic microflora profile, bowel function, and blood cholesterol levels in constipated elderly people--a placebo-controlled, diet-controlled trial. Nutrition. 2011 Apr;27(4):445-50. doi: 10.1016/j.nut.2010.05.012. Epub 2010 Jul 10. PMID 20624673
- [Background] Davis LM, Martinez I, Walter J, Hutkins R. A dose dependent impact of prebiotic galactooligosaccharides on the intestinal microbiota of healthy adults. Int J Food Microbiol. 2010 Dec 15;144(2):285-92. doi: 10.1016/j.ijfoodmicro.2010.10.007. Epub 2010 Oct 14. PMID 21059476
- [Background] Komanduri S, Gillevet PM, Sikaroodi M, Mutlu E, Keshavarzian A. Dysbiosis in pouchitis: evidence of unique microfloral patterns in pouch inflammation. Clin Gastroenterol Hepatol. 2007 Mar;5(3):352-60. doi: 10.1016/j.cgh.2007.01.001. PMID 17368235